CLINICAL TRIAL: NCT06571331
Title: A Randomized, Double Blind, Placebo-controlled, Parallel Arm Clinical Trial of De-Stress and Snooze Gummies in Reducing Stress, Insomnia Disorder, Associated Symptoms and Overall Quality of Life
Brief Title: A Clinical Trial of De-Stress & Snooze Gummies in Reducing Stress and Insomnia Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Herbolab India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MHC/CT/24-25/019; CTRI/2024/07/071253 (Registry Identifier: Clinical trials registry of India)
Record Dates: First submitted 2024-08-10; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Stress; Insomnia; Quality of Life
Keywords: Stress; Insomnia; Quality of Life
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, Double Blind, Parallel Group, Placebo-Controlled Trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- De-Stress & Snooze Gummies-U001 (Experimental)
  Interventions: Other: De-Stress & Snooze Gummies-U001
- De-Stress & Snooze Gummies-I001 (Experimental)
  Interventions: Other: De-Stress & Snooze Gummies-I001
- Placebo Gummies 002 (Placebo Comparator)
  Interventions: Other: Placebo Gummies 002

INTERVENTIONS:
Other: De-Stress & Snooze Gummies-U001 — Two gummies daily in sequence 30-45 minutes before bed for 60 days
  Arms: De-Stress & Snooze Gummies-U001
Other: De-Stress & Snooze Gummies-I001 — Two gummies daily in sequence 30-45 minutes before bed for 60 days
  Arms: De-Stress & Snooze Gummies-I001
Other: Placebo Gummies 002 — Two gummies daily in sequence 30-45 minutes before bed for 60 days
  Arms: Placebo Gummies 002

SUMMARY:
The current study focuses on clinical validation of efficacy of nutraceutical product in management of sleep disorder. Improved sleep quality contributes significantly to cognitive function. With a good night's sleep, individuals often find themselves more alert, focused, and better equipped to handle complex tasks and problem-solving scenarios. This can enhance productivity at work, as well as improve the ability to engage in meaningful conversations and activities. Memory consolidation, which occurs during sleep, is also optimized, leading to better retention of information and a sharper mind.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial of De-Stress and Snooze Gummies in reducing stress, insomnia disorder, associated symptoms, and overall quality of life.

More than 60 Participants will be randomized to either one of the following groups:

Group A, Group B, and Group C will involve 20 participants each group (1:1:1 ratio) will be advised to take Destress and snooze gummies - U001, Destress and snooze gummies - I001, and Placebo gummies-002, respectively two gummies in sequence daily, 30 minutes before bed, for 60 days. The treatment duration is of 60 days and the study duration is of 68 days. The efficacy of the investigational product will be compared between the groups.

Concomitant diseases/medication assessment will be performed on screening.

Assessments of changes in stress through PSS scores, serum serotonin, restorative sleep by RSQ-W score, under eye dark circles based on bespoke scale, and headache by VAS score will be conducted on screening, day 30 and day 60.

Changes in serum cortisol levels will be evaluated at screening, day 15, and day 60. Additionally, participants' sleep diaries will be assessed to determine the changes in total sleep time, sleep latency, number of awakenings, wake time after sleep onset, sleep efficiency (total sleep time/time in bed * 100), and levels of alertness and drowsiness and actigraphy assessment using Fitbit device to evaluate sleep efficiency (deep sleep, light sleep, and REM sleep duration, as well as overall sleep scores) which will be tracked for 10 individuals (3-4 subjects per group) at baseline, day 30, and day 60.

Changes in the Functional Outcomes of Sleep Questionnaire (FOSQ-10) and the abbreviated Profile of Mood States (POMS-A) score to investigate mood changes and safety through complete blood count, liver function test, and kidney function test will be assessed at screening and day 60.

Changes in the modified sleep regularity and medication withdrawal questionnaire (MSRMWQ) score will be assessed after ceasing treatment for one week (day 68), telephonically.

Treatment compliance and tolerability will be assessed at day 30 and day 60, and safety of the investigational treatment in terms of adverse events will be assessed at baseline, day 15, day 45, and day 60. Changes in vital sign parameters will be assessed at screening, baseline, day 15, day 30, day 45 and day 60.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 21-50 years both inclusive
2. Suffering from self-reported mild to moderate stress on the PSS scale score less than or equal to 26
3. Participants willing to participate in clinical trials and who have read understood and signed the informed consent form
4. Participants diagnosed with insomnia disorder based on the Diagnostic and Statistical Manual of Mental Disorders text revision DSM-V-TR
5. Insomnia Severity Index more than 7 and less than 21 i.e. mild to moderate
6. Participants with a diagnosis of mild or moderate depression patient's health questionnaire PHQ-9 score of less than or equal to 14
7. Participants with a diagnosis of mild or moderate generalized anxiety disorder GAD -7 questionnaire score of less than or equal to 10.

Exclusion Criteria:

1. Difficulty sleeping due to a medical condition
2. History of a neurological disorder
3. History of bipolar disorder psychotic disorder or posttraumatic stress disorder or current psychiatric disorder that requires medication
4. On-going depression and generalized anxiety disorder diagnosis on PHQ 9 score greater than or equal to 15 and GAD-7 score greater than or equal to 11 scales
5. History of substance abuse or dependence
6. History or current evidence of a clinically significant cardiovascular disorder at pre-study visit
7. Taking certain prohibited medications
8. Consumption of greater than 10 cigarettes a day
9. Participants who consume greater than or equal to 120 mg/day of caffeine and are unwilling to restrict their intake throughout the study
10. Current evidence or history of malignancy less than or equal to 5 years prior to signing informed consent
11. Participants currently using any nutraceutical, allopathic, or ayurvedic supplement for stress or insomnia management
12. Known hypersensitivity to any ingredients of product
13. Pregnant or lactating women, as well as women of childbearing potential who are not using contraception or intending to conceive during the study
14. Other conditions, which in the opinion of the investigators, makes the participant unsuitable for enrolment or could interfere with his her participation in and completion of the protocol.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | Screening, day 30 and day 60
  The PSS-10 is widely used for measuring psychological distress. It contains 10 questions on a five-point scale from 0 to 4. The higher the score, the greater the feeling of stress. PSS-10 Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Restorative Sleep Questionnaire Weekly Version (RSQ-W) | Screening, day 30 and day 60
  Total score of how an individual rates the restorative value of his/her sleep in the morning using the weekly version of the Restorative Sleep Questionnaire (RSQ-Weekly). It is a 9 item scale questioner. Scoring interpretation: A total score is calculated as the average of the questionnaire items. The total score ranges from 0 to 100, with higher scores indicating better restorative sleep. To convert the average score to a 0-100 scale, the following transformation is used: RSQ-W Total Score = {RSQ-W Average Score Across Completed Items - 1} *25.
Number of Participants Who Showed Improvement in Under Eye Dark Circle | Screening, day 30 and day 60
  The interpretation will be like No Dark Circles (No visible dark circles under the eyes); 1: Minimal Dark Circles (Slight discoloration or shadow, barely noticeable); 2: Mild Dark Circles (Noticeable darkening, but not prominent or severe); 3: Moderate Dark Circles (Prominent dark circles with moderate intensity); 4: Severe Dark Circles (Intense and distinct dark circles, may appear blueish-black); 5: Blueish Black Dark Circles (Extreme and prominent dark circles with a deep blue or black hue).
visual analogue scale | Screening, day 30 and day 60
  Visual analogue scale score- for evaluation of fatigue, nausea, palpitation, breathlessness A higher score (10) represents severe symptoms and a lower score (0) represents no symptoms.
Change in Sleep Efficiency | Baseline, day 30 ad day 60
  Sleep efficiency will be calculated using information by actigraphy from Fitbit device.
  Sleep efficiency in terms of - Deep sleep, light sleep, REM sleep duration and overall sleep score by actigraphy (Fitbit device) for 10 subjects (3-4 subjects in each group).
Changes in Modified sleep regularity and medication withdrawal questionnaire (MSRMWQ) | Score after stopping treatment for 1 week (day 68)
  The Modified Sleep Regularity and Medication Withdrawal Questionnaire (MSRMWQ) is a tool designed to assess changes in sleep patterns and the impact of medication withdrawal on sleep. Total score categories: Part I 00-10 = Poor sleep regularity 21-30 = Better sleep regularity 11-20 = Good sleep regularity 31-40 = Excellent sleep regularity Parameter-wise scoring by 4 point Linkert scale: Part II 0 = No symptom 1 = Resolved symptom 2 = Ongoing symptoms requiring no medical assistance 3 = Ongoing symptoms requiring medical assistance
Changes in serum cortisol levels | Screening, day 15 and day 60
  The cortisol secretion will be evaluated by measuring morning serum cortisol levels.
Change in serum serotonin levels | Screening, day 30 and day 45
  The serotonin secretion will be evaluated by measuring morning serum serotonin levels.
Change in FOSQ-10 score Profile of Mood State (POMS) questionnaire | Screening and day 28
  Functional Outcomes of Sleep Questionnaire (FOSQ-10): Subscale scores range from 1-4 (1= extreme difficulty, 2= moderate difficulty, 3= a little difficulty, 4= no difficulty) with total scores ranging from 10-40 with higher scores indicating higher functional.
Profile of Mood State (POMS) questionnaire | Screening and day 28
  The Profile of Mood States (POMS) is a widely used instrument that measures mood using a 40 item questionnaire with each item rated using a response scale of five categories ranging from "not at all" to "Extremely". Higher score indicates worse mood. Total POMS score categories and stress inference:
  0-40 = A little; 81-120= Quite a lot; 41-80= Moderately; 121-160= extremely.
Changes in outcomes from participant sleep diary | Baseline, day 30 and day 60
  Sleep diary parameters - total sleep time in minutes, sleep latency in minutes, number of awakenings in numbers, wake time after sleep onset in minutes, sleep efficiency in percentage (Total sleep time/ time in bed*100), alertness and drowsiness will be recorded using 5-point scale.

SECONDARY OUTCOMES:
Safety of participant Assessed using adverse events | Screening, baseline, day 15, day 30, day 45, day 60
  It is measured in terms of No. of events
Safety of participant Assessed using treatment compliance and tolerability of investigational product | Screening, baseline, day 15, day 30, day 45, day 60
  It is measure in terms of percentage
Systolic blood pressure difference from reference measurement (mmHg) | Screening and day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Diastolic blood pressure difference from reference measurement (mmHg) | Screening and day 60
  Assessed against standard clinical grade instrument: automated oscillometric blood pressure device (mmHg)
Pulse rate difference from reference measurement (beats per minute) | Screening and day 60
  Assessed against standard clinical grade instrument: Finger-based pulse oximeter (beats per minute)
Complete blood count | Screening and day 60
  White blood cell and platelet count [Thousand per microliter (Thousand/uL)] Red blood cell count [Millions per microliter (million/uL)]
Serum Glutamic Pyruvic Transaminase (SGPT) | Screening and day 60
  Blood level of SGPT was measured. (U/L)
serum glutamic-oxaloacetic transaminase (SGOT) | Screening and day 60
  Blood level of SGOT was measured. (U/L)
Creatinine | Screening and day 60
  Creatinine difference from reference measurement (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ramshyam Agarwal, MBBS, DNB, Principal Investigator — Lokmanya Medical Research Centre and Hospital

IPD SHARING:
Plan to Share IPD: No